CLINICAL TRIAL: NCT06233942
Title: Phase 1a/1b Study of BG-C9074, an Antibody Drug Conjugate Targeting B7H4, as Monotherapy and in Combination With Other Anticancer Therapies in Patients With Advanced Solid Tumors
Brief Title: Phase 1a/1b First-in-Human Study of BG-C9074 Alone and in Combination With Other Anticancer Therapies in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG-C9074-101
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor
Keywords: BG-C9074; Tislelizumab; Advanced Solid Tumors; first-in-human; B7H4
MeSH Terms: interventions — tislelizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Phase 1a: Part A (Monotherapy Dose Escalation) (Experimental): BG-C9074 monotherapy dose escalation
  Interventions: Drug: BG-C9074
- Phase 1a: Part B (Monotherapy Safety Expansion) (Experimental): BG-C9074 dose levels that have been determined to be safe and tolerable in Part A will be investigated.
  Interventions: Drug: BG-C9074
- Phase 1a: Part C (Combination Therapy Dose Escalation) (Experimental): BG-C9074 plus tislelizumab combination at the recommended dose for expansion (RDFE).
  Interventions: Drug: BG-C9074; Drug: Tislelizumab
- Phase 1a: Part D (Japan Cohort) (Experimental): A separate cohort in Japan will evaluate the safety of BG-C9074 monotherapy in Japanese participants with select solid tumors
  Interventions: Drug: BG-C9074
- Phase 1b: Monotherapy Dose Expansion (Experimental): The monotherapy dose expansion phase will begin once the BG-C9074 monotherapy RDFE and dosing schedule have been determined from Parts A and B in Phase 1a.
  Interventions: Drug: BG-C9074
- Phase 1b: Combination Therapy Dose Expansion (BG-C9074 plus tislelizumab) (Experimental): This arm will assess BG-C9074 plus tislelizumab as first-line therapy in select solid tumors after completion of the dose escalation phase.
  Interventions: Drug: BG-C9074; Drug: Tislelizumab
- Phase 1b: Combination Therapy Dose Expansion (BG-C9074 plus bevacizumab) (Experimental): This arm will assess BG-C9074 plus bevacizumab in select solid tumors participants after establishing the recommended monotherapy dose and schedule.
  Interventions: Drug: BG-C9074; Drug: Bevacizumab

INTERVENTIONS:
Drug: BG-C9074 — administered by intravenous infusion
Drug: Tislelizumab — administered by intravenous infusion
  Arms: Phase 1a: Part C (Combination Therapy Dose Escalation); Phase 1b: Combination Therapy Dose Expansion (BG-C9074 plus tislelizumab)
Drug: Bevacizumab — administered by intravenous infusion
  Arms: Phase 1b: Combination Therapy Dose Expansion (BG-C9074 plus bevacizumab)

SUMMARY:
This is a first-in-human, dose finding and dose expansion study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of BG-C9074 alone and in combination with other anticancer therapies in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide a signed and dated written informed consent prior to any study-specific procedures, sampling, or data collection.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
3. Participants with selected histologically or cytologically confirmed advanced, metastatic, and unresectable solid tumors who have previously received standard systemic therapy and whose cancer is not amenable to therapy with curative intent, and for whom further treatment is not available or not tolerated. Enrollment will be limited to participants with hormone receptor-positive/human epidermal growth factor receptor 2-negative (HR+/HER2-) breast cancer, cholangiocarcinoma (CCA), endometrial cancer, squamous non-small cell lung cancer (NSCLC), triple-negative breast cancer (TNBC), or ovarian cancer. Enrollment in the Japan cohort will be limited to participants with HR+/HER2- breast cancer, TNBC, endometrial cancer, or ovarian cancer.
4. ≥ 1 measurable lesion per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1)
5. Able to provide an archived tumor tissue sample.
6. Adequate bone marrow and organ function.
7. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and for ≥ 7 months after the last dose of study drug(s).
8. Nonsterile males must be willing to use a highly effective method of birth control for the duration of the study treatment period and for ≥ 4 months after the last dose of study drug(s).

Exclusion Criteria:

1. Prior treatment with a B7 homolog 4 (B7H4)-targeting antibody-drug conjugate (ADC) or an ADC with a topoisomerase 1 inhibitor (TOP1i) payload.
2. Active leptomeningeal disease or uncontrolled, untreated brain metastasis
3. Any malignancy ≤ 2 years before the first dose of study treatment(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast).
4. History of interstitial lung disease, ≥ Grade 2 noninfectious pneumonitis, oxygen saturation at rest < 92%, or requirement for supplemental oxygen (including intermittent use) at baseline.
5. Uncontrolled diabetes.
6. Infection (including tuberculosis infection) requiring systemic (oral or intravenous) antibacterial, antifungal, or antiviral therapy ≤ 14 days before the first dose of study treatment(s).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2027-09-28 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 3 years
  Number of participants with AEs and SAEs (as graded by the National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] Version [v] 5.0),, including findings from physical examinations, electrocardiograms (ECGs), laboratory assessments, and that meet protocol-defined dose-limiting toxicity criteria.
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BG-C9074 | Approximately 18 months
  Defined as the highest dose evaluated for which the estimated toxicity rate is closest to the target toxicity rate of 28% or the highest dose administered, respectively
Phase 1a: Recommended Dose for Expansion (RDFE) of BG-C9074. | Approximately 18 months
  The potential RDFE(s) of BG-C9074 alone and in combination with tislelizumab will be determined based on the MTD or MAD, taking into consideration the long-term tolerability, PK, pharmacodynamics, preliminary antitumor activity, and any other relevant data, as available
Phase 1b: Overall Response Rate (ORR) as monotherapy and in combination with tislelizumab | Approximately 3 years
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) assessed by the investigator using RECIST v1.1.
Phase 1b: Recommended Phase 2 dose (RP2D) of BG-C9074 as monotherapy and in combination with bevacizumab or tislelizumab | Approximately 30 months
  The RP2D of BG-C9074 will be determined based on safety, PK, pharmacodynamics, preliminary antitumor activity, and other relevant data, as available.

SECONDARY OUTCOMES:
Phase 1a: ORR as monotherapy and in combination with tislelizumab | Approximately 3 years
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) assessed by the investigator using RECIST v1.1.
Phase 1b: ORR as monotherapy and in combination with bevacizumab or tislelizumab | Approximately 3 years
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) assessed by the investigator using RECIST v1.1.
Phase 1b: ORR per B7-H4 (B7 homolog 4) protein expression | Approximately 3 years
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) assessed by the investigator using RECIST v1.1 and evaluated according to the amount of B7-H4 (B7 homolog 4) protein expressed in their tumors
Duration of Response (DOR) | Approximately 3 years
  Duration of response (DOR) is defined as the time from the first determination of an objective response per RECIST v1.1 until the first documentation of disease progression or death, whichever occurs first, as assessed by the investigator
Duration of Response (DOR) per B7-H4 protein expression | Approximately 3 years
  Duration of response (DOR) is defined as the time from the first determination of an objective response per RECIST v1.1 until the first documentation of disease progression or death, whichever occurs first, as assessed by the investigator, and evaluated according to the amount of B7-H4 protein expressed in the tumors
Disease Control Rate (DCR) | Approximately 3 years
  DCR is defined as the percentage of participants with best overall response of CR, PR, or stable disease, as assessed by the investigator
Disease Control Rate (DCR) per B7-H4 protein expression | Approximately 3 years
  DCR is defined as the percentage of participants with best overall response of CR, PR, or stable disease, as assessed by the investigator, and evaluated according to the amount of B7-H4 protein expressed in the tumors
Clinical Benefit Rate (CBR) | Approximately 3 years
  CBR is defined as the percentage of participants with best overall response of confirmed CR, PR, or stable disease lasting ≥ 24 weeks as assessed by investigator.
Clinical Benefit Rate (CBR) per B7-H4 protein expression | Approximately 3 years
  CBR is defined as the percentage of participants with best overall response of confirmed CR, PR, or stable disease lasting ≥ 24 weeks as assessed by investigato, and evaluated according to the amount of B7-H4 protein expressed in the tumors
Phase 1b: Progression Free Survival (PFS) | Approximately 3 years
  PFS is defined as the time from the date of the first dose of study drug(s) to the date of the first documentation of progressive disease assessed by the investigator using RECIST v1.1 or death, whichever occurs first.
Phase 1b: Number of Participants with AEs and SAEs | Approximately 3 years
  Number of participants with AEs and SAEs, including findings from physical examinations, electrocardiograms (ECGs), and laboratory assessments.
Maximum observed plasma concentration (Cmax) for BG-C9074 | Twice in the first four months
Minimum observed plasma concentration (Cmin) for BG-C9074 | Approximately 3 years
Time to reach maximum observed plasma concentration (Tmax) for BG-C9074 | Twice in the first four months
Half-life (t1/2) for BG-C9074 | Twice in the first four months
Area under the concentration-time curve (AUC) for BG-C9074 | Twice in the first four months
Apparent clearance (CL/F) for BG-C9074 | Twice in the first four months
Apparent volume of distribution (Vz/F) for BG-C9074 | Twice in the first four months
Accumulation ratio for BG-C9074 | Twice in the first four months
Plasma concentrations for BG-C9074 | Approximately 3 years
Phase 1a: Number of participants with anti-drug antibodies (ADAs) to BG-C9074 and tislelizumab | Approximately 3 years
Phase 1b: Number of participants with anti-drug antibodies (ADAs) to BG-C9074 | Approximately 3 years
Serum concentration of BG-C0974 | Approximately 3 years
Serum concentration of Tislelizumab | Approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (27):
- United States (5):
  - Usc Norris Comprehensive Cancer Center (Nccc), Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Florida Cancer Specialist Research Institute Lake Nona, Orlando, Florida
  - Sidney Kimmel Comprehensive Cancer At Johns Hopkins, Baltimore, Maryland
  - James Cancer Hospital and Solove Research Institute, Columbus, Ohio
- Australia (8):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Cancer Care Wollongong, Wollongong, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Health, Clayton, Victoria
  - Cabrini Hospital Malvern, Malvern East, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (14):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/